CLINICAL TRIAL: NCT06322446
Title: Effects of a Strength Exercise Program on Muscular Health in People With CF Treated With Modulators of the Cystic Fibrosis Transmembrane Conductance Regulator Receptor (CFTR)
Brief Title: Exercise in People With Cystic Fibrosis on CFTR Modulator Therapy
Acronym: FIQMODE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Collaborators: Carlos III Health Institute (Other Government); Universidad Europea de Madrid (Other); Hospital Universitario La Paz (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Responsible Party: Principal Investigator, Margarita Pérez-Ruiz, full professor in Physical Activity and Health, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI23/00299
Record Dates: First submitted 2024-02-22; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis
Keywords: Physical Fitness; Muscle Strength; Resistance Training; Lung funcion
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Telematic Exercise:
  A remotely supervised resistance exercise program will be carried out for 16 weeks, with two weekly sessions lasting approximately 60 minutes each. Training will be performed in groups of four patients, according to their lung function/physical fitness.
  The first training session will be on site (University) for familiarization, planning and adjustment of the exercises, and the following sessions will be performed online. Each session is divided into: (i) Warm-up and joint mobility; (ii) main part: strength exercises for different muscle groups; and (iii) cool down: stretching and breathing exercises.
  Interventions: Other: Exercise
- Control (No Intervention): Control group will follow routine recommendations from the multidisciplinary CF team based on WHO´s guidelines

INTERVENTIONS:
Other: Exercise — 16-week exercise intervention: At the beginning of the intervention, we will conduct a face-to-face familiarisation session with the exercises of the training programme. The intervention will consist of 2 sessions/week for 16 weeks. Each session consists of three stages: (i) Warm-up: 10 min of joint mobility and low intensity exercises involving the musculature to be worked in that session; (ii) Main part: circuit training mainly composed of strength exercises targeting the different muscle groups of the body and playing activities (iii) Cool down: 10 min with guided breathing work and stretching of the main muscle groups worked
  Arms: Intervention

SUMMARY:
Recently, the treatment of Cystic Fibrosis (CF) incorporated new modulators/enhancers of the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR). It is thus increasingly important to study the side effects of these drugs, their extrapulmonary effects and possible interaction with other drugs and with exercise. For this purpose, a randomized controlled trial is proposed to determine the effects of a telematic exercise intervention on muscle health, in a group of 48 children and adolescents with CF treated with these new generation CFTR modulators. They will be randomly assigned to two groups (exercise and control group). The effect of the intervention will be analysed measuring the variables of muscle health, cardiorespiratory fitness, lung function, body composition, inflammatory biomarkers and miRNAs. After completion of the intervention program, adherence to exercise and clinical evolution after one year will be analysed.

DETAILED DESCRIPTION:
Specific objectives

1. To determine the effects of a strength exercise intervention in a group of children and adolescents with cystic fibrosis treated with new generation CFTR modulators on: (1.i) peripheral muscle strength; (1.ii) respiratory muscle strength; (1.iii) muscle mass and (1.iv) biomarkers of muscle damage.
2. To determine the effects of a strength exercise intervention in a group of children and adolescents with cystic fibrosis being treated with new generation CFTR modulators on: (2.i) cardiorespiratory fitness; (2.ii) body composition and (2.iii) lung function.
3. To determine the effects of a strength-based exercise intervention in a group of children and adolescents with cystic fibrosis treated with new-generation CFTR modulators on: (3.i) biomarkers of inflammatory status and (3.ii) expression of associated miRNAs.
4. To determine the effects of a strength-based exercise intervention in a group of children and adolescents with cystic fibrosis treated with the new generation CFTR modulators on the levels of Elexaxcaftor/Ivacaftor/Tezacaftor and their metabolites.
5. To assess the clinical evolution and adherence to exercise after 6 months of the programme in children and adolescents with cystic fibrosis treated with the new generation of CFTR modulators.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with CF.
* patients between 6-20 years of age.
* patients receiving treatment with new CFTR protein modulating medication
* reading, acceptance and signing of the informed consent form.

Exclusion Criteria:

* CF patients with symptoms of pulmonary exacerbation during the last four weeks.
* with a diagnosis of other cardiorespiratory lung diseases progressing to a symptom of persistent respiratory dysfunction.
* CF patients with musculoskeletal alterations that influence assessments.
* CF patient who is pregnant during the time of the study
* CF patient with cognitive impairment;
* CF patient with incomplete dosing of modulator therapy;

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Changes in peripheral muscle strength | Baseline, pre-intervention and immediately after the intervention.
  Upper and lower limbs muscle strength (kg) will be evaluated using dynamometers.
Changes in inspiratory/expiratory muscle strength (MIP/MEP) (cmH2O) | Baseline, pre-intervention and immediately after the intervention
  Inspiratory and expiratory muscle strength: maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured.
Changes in functional capacity: lower limbs power capacity | Baseline, pre-intervention and immediately after the intervention
  30 seconds sit-to-stand test. Unit of measurement: number of repetitions.
Changes in functional capacity: walking capacity | Baseline, pre-intervention and immediately after the intervention
  10m Time (s) Up and Go tests.
Change in Cardiorespiratory fitness: maximal oxygen consumption | Baseline, pre-intervention and immediately after the intervention
  To assess cardiorespiratory fitness, a treadmill and a gas analyser will be used. The test aims to determine maximal oxygen consumption (VO2peak in ml/kg/min). VO2peak will be recorded as the highest value obtained during a continuous 30 s period.
Change in Cardiorespiratory fitness: Ventilatory threshold VT1 | Baseline, pre-intervention and immediately after the intervention
  To assess cardiorespiratory fitness, a treadmill and a gas analyser will be used. The test aims to determine the ventilatory threshold VT1 in response to maximal effort. VT1 will be determined using the criteria of an increase in both ventilatory equivalent for oxygen consumption (VE/VO2) and end-tidal oxygen pressure without an increase in ventilatory equivalent for carbon dioxide production (VE/VCO2).

SECONDARY OUTCOMES:
Changes in Pulmonary Function: forced vital capacity (FVC) | Baseline, pre-intervention and immediately after the intervention
  Spirometry will assess: forced vital capacity (FVC) in milliliters and percentage of predicted value
Changes in Pulmonary Function: Forced expiratory volume in the first second (FEV1) | Baseline, pre-intervention and immediately after the intervention
  Spirometry will assess: forced expiratory volume in the first second (FEV1).Data will be expressed in absolute values and z-score based on the Global Lung Initiative (GLI) reference equation establishing as a limit of normality (LIN) a z-score value for FEV1 between -1.64 and + 1.64.
Changes in the anthropometric and body composition: Weight | Baseline, pre-intervention and immediately after the intervention
  Weight (kg)
Changes in the anthropometric and body composition: Height | Baseline, pre-intervention and immediately after the intervention
  Height (cm)
Changes in the anthropometric and body composition: BMI | Baseline, pre-intervention and immediately after the intervention
  BMI (kg/m2)
Changes in body composition: Total fat mass | Baseline, pre-intervention and immediately after the intervention
  Total fat mass (kg)
Changes in body composition: FMI | Baseline, pre-intervention and immediately after the intervention
  fat mass index (FMI) (kg/m2),
Changes in body composition: lean mass kg | Baseline, pre-intervention and immediately after the intervention
  Lean mass in kg
Changes in body composition: lean mass % | Baseline, pre-intervention and immediately after the intervention
  Lean mass in %
Changes in quality of life using the Cystic Fibrosis Questionnaire | Baseline, pre-intervention and immediately after the intervention
  Scores range from 0 to 100 with higher scores corresponding to better quality of life.
Changes in plasma levels muscle damage biomarkers | Baseline, pre-intervention and immediately after the intervention
  Blood levels biomarkers of muscle damage as CK measured in micrograms per litre (mcg/L)
Changes in plasma levels of inflammation: hs-CRP | Baseline, pre-intervention and immediately after the intervention
  High-sensitivity C-reactive protein (hs-CRP) assay in milligrams/litre
Changes in plasma levels of inflammation: Interleukins | Baseline, pre-intervention and immediately after the intervention
  Analysis of interleukins such as IL6, IL-10 in picograms/millilitre

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Perez Ruiz, PhD, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Facultad de Ciencias de la Actividad Física y Deporte - INEF UPM, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bell SC, Mall MA, Gutierrez H, Macek M, Madge S, Davies JC, Burgel PR, Tullis E, Castanos C, Castellani C, Byrnes CA, Cathcart F, Chotirmall SH, Cosgriff R, Eichler I, Fajac I, Goss CH, Drevinek P, Farrell PM, Gravelle AM, Havermans T, Mayer-Hamblett N, Kashirskaya N, Kerem E, Mathew JL, McKone EF, Naehrlich L, Nasr SZ, Oates GR, O'Neill C, Pypops U, Raraigh KS, Rowe SM, Southern KW, Sivam S, Stephenson AL, Zampoli M, Ratjen F. The future of cystic fibrosis care: a global perspective. Lancet Respir Med. 2020 Jan;8(1):65-124. doi: 10.1016/S2213-2600(19)30337-6. Epub 2019 Sep 27. PMID 31570318
- [Background] Kerem B, Rommens JM, Buchanan JA, Markiewicz D, Cox TK, Chakravarti A, Buchwald M, Tsui LC. Identification of the cystic fibrosis gene: genetic analysis. Science. 1989 Sep 8;245(4922):1073-80. doi: 10.1126/science.2570460.
- [Background] Riordan JR, Rommens JM, Kerem B, Alon N, Rozmahel R, Grzelczak Z, Zielenski J, Lok S, Plavsic N, Chou JL, et al. Identification of the cystic fibrosis gene: cloning and characterization of complementary DNA. Science. 1989 Sep 8;245(4922):1066-73. doi: 10.1126/science.2475911.
- [Background] Rommens JM, Zengerling-Lentes S, Kerem B, Melmer G, Buchwald M, Tsui LC. Physical localization of two DNA markers closely linked to the cystic fibrosis locus by pulsed-field gel electrophoresis. Am J Hum Genet. 1989 Dec;45(6):932-41. PMID 2589321
- [Background] Elborn JS. Cystic fibrosis. Lancet. 2016 Nov 19;388(10059):2519-2531. doi: 10.1016/S0140-6736(16)00576-6. Epub 2016 Apr 29. PMID 27140670
- [Background] Bergeron C, Cantin AM. Cystic Fibrosis: Pathophysiology of Lung Disease. Semin Respir Crit Care Med. 2019 Dec;40(6):715-726. doi: 10.1055/s-0039-1694021. Epub 2019 Oct 28. PMID 31659725
- [Background] Singh VK, Schwarzenberg SJ. Pancreatic insufficiency in Cystic Fibrosis. J Cyst Fibros. 2017 Nov;16 Suppl 2:S70-S78. doi: 10.1016/j.jcf.2017.06.011. PMID 28986019
- [Background] Kamal N, Surana P, Koh C. Liver disease in patients with cystic fibrosis. Curr Opin Gastroenterol. 2018 May;34(3):146-151. doi: 10.1097/MOG.0000000000000432. PMID 29438119
- [Background] Ratchford TL, Teckman JH, Patel DR. Gastrointestinal pathophysiology and nutrition in cystic fibrosis. Expert Rev Gastroenterol Hepatol. 2018 Sep;12(9):853-862. doi: 10.1080/17474124.2018.1502663. Epub 2018 Aug 3. PMID 30019967
- [Background] Quinton PM. Cystic fibrosis: lessons from the sweat gland. Physiology (Bethesda). 2007 Jun;22:212-25. doi: 10.1152/physiol.00041.2006. PMID 17557942
- [Background] Shteinberg M, Taylor-Cousar JL, Durieu I, Cohen-Cymberknoh M. Fertility and Pregnancy in Cystic Fibrosis. Chest. 2021 Dec;160(6):2051-2060. doi: 10.1016/j.chest.2021.07.024. Epub 2021 Jul 18. PMID 34284004
- [Background] Reznikov LR. Cystic Fibrosis and the Nervous System. Chest. 2017 May;151(5):1147-1155. doi: 10.1016/j.chest.2016.11.009. Epub 2016 Nov 19. PMID 27876591
- [Background] Khalaf M, Scott-Ward T, Causer A, Saynor Z, Shepherd A, Gorecki D, Lewis A, Laight D, Shute J. Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) in Human Lung Microvascular Endothelial Cells Controls Oxidative Stress, Reactive Oxygen-Mediated Cell Signaling and Inflammatory Responses. Front Physiol. 2020 Jul 29;11:879. doi: 10.3389/fphys.2020.00879. eCollection 2020. PMID 32848840
- [Background] Tousson A, Van Tine BA, Naren AP, Shaw GM, Schwiebert LM. Characterization of CFTR expression and chloride channel activity in human endothelia. Am J Physiol. 1998 Dec;275(6):C1555-64. doi: 10.1152/ajpcell.1998.275.6.C1555. PMID 9843717
- [Background] Plebani R, Tripaldi R, Lanuti P, Recchiuti A, Patruno S, Di Silvestre S, Simeone P, Anile M, Venuta F, Prioletta M, Mucilli F, Del Porto P, Marchisio M, Pandolfi A, Romano M. Establishment and long-term culture of human cystic fibrosis endothelial cells. Lab Invest. 2017 Nov;97(11):1375-1384. doi: 10.1038/labinvest.2017.74. Epub 2017 Jul 31. PMID 28759010
- [Background] Totani L, Plebani R, Piccoli A, Di Silvestre S, Lanuti P, Recchiuti A, Cianci E, Dell'Elba G, Sacchetti S, Patruno S, Guarnieri S, Mariggio MA, Mari VC, Anile M, Venuta F, Del Porto P, Moretti P, Prioletta M, Mucilli F, Marchisio M, Pandolfi A, Evangelista V, Romano M. Mechanisms of endothelial cell dysfunction in cystic fibrosis. Biochim Biophys Acta Mol Basis Dis. 2017 Dec;1863(12):3243-3253. doi: 10.1016/j.bbadis.2017.08.011. Epub 2017 Aug 25. PMID 28847515
- [Background] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Shazam Hussain M, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. Int J Stroke. 2018 Aug;13(6):612-632. doi: 10.1177/1747493018778713. Epub 2018 May 22. No abstract available. PMID 29786478
- [Background] Calella P, Valerio G, Brodlie M, Donini LM, Siervo M. Cystic fibrosis, body composition, and health outcomes: a systematic review. Nutrition. 2018 Nov;55-56:131-139. doi: 10.1016/j.nut.2018.03.052. Epub 2018 Apr 6. PMID 29981489
- [Background] Galluzzi L, Kroemer G. Etiological involvement of CFTR in apparently unrelated human diseases. Mol Cell Oncol. 2018 Dec 27;6(1):1558874. doi: 10.1080/23723556.2018.1558874. eCollection 2019. No abstract available. PMID 30788425
- [Background] Zemanick ET, Ong T, Daines CL, Dellon EP, Muhlebach MS, Esther CR Jr. Highlights from the 2015 North American Cystic Fibrosis Conference. Pediatr Pulmonol. 2016 Jun;51(6):650-7. doi: 10.1002/ppul.23441. Epub 2016 Apr 13. PMID 27074261
- [Background] Angelis A, Kanavos P, Lopez-Bastida J, Linertova R, Nicod E, Serrano-Aguilar P; BURQOL-RD Research Network. Social and economic costs and health-related quality of life in non-institutionalised patients with cystic fibrosis in the United Kingdom. BMC Health Serv Res. 2015 Sep 28;15:428. doi: 10.1186/s12913-015-1061-3. PMID 26416027
- [Background] Nichols DP, Donaldson SH, Frederick CA, Freedman SD, Gelfond D, Hoffman LR, Kelly A, Narkewicz MR, Pittman JE, Ratjen F, Sagel SD, Rosenfeld M, Schwarzenberg SJ, Singh PK, Solomon GM, Stalvey MS, Kirby S, VanDalfsen JM, Clancy JP, Rowe SM. PROMISE: Working with the CF community to understand emerging clinical and research needs for those treated with highly effective CFTR modulator therapy. J Cyst Fibros. 2021 Mar;20(2):205-212. doi: 10.1016/j.jcf.2021.02.003. Epub 2021 Feb 19. PMID 33619012
- [Background] Burgener EB, Moss RB. Cystic fibrosis transmembrane conductance regulator modulators: precision medicine in cystic fibrosis. Curr Opin Pediatr. 2018 Jun;30(3):372-377. doi: 10.1097/MOP.0000000000000627. PMID 29538046
- [Background] Gramegna A, Contarini M, Aliberti S, Casciaro R, Blasi F, Castellani C. From Ivacaftor to Triple Combination: A Systematic Review of Efficacy and Safety of CFTR Modulators in People with Cystic Fibrosis. Int J Mol Sci. 2020 Aug 16;21(16):5882. doi: 10.3390/ijms21165882. PMID 32824306
- [Background] Elborn JS. Adult Care in Cystic Fibrosis. Semin Respir Crit Care Med. 2019 Dec;40(6):857-868. doi: 10.1055/s-0039-3400289. Epub 2019 Dec 30. PMID 31887770
- [Background] Williams CA, Barker AR, Denford S, van Beurden SB, Bianchim MS, Caterini JE, Cox NS, Mackintosh KA, McNarry MA, Rand S, Schneiderman JE, Wells GD, Anderson P, Beever D, Beverley Z, Buckley R, Button B, Causer AJ, Curran M, Dwyer TJ, Gordon W, Gruet M, Harris RA, Hatziagorou E, Erik Hulzebos HJ, Kampouras A, Morrison L, Camara MN, Reilly CM, Sawyer A, Saynor ZL, Shelley J, Spencer G, Stanford GE, Urquhart DS, Young R, Tomlinson OW; Youth Activity Unlimited - A Strategic Research Centre of the UK Cystic Fibrosis Trust. The Exeter Activity Unlimited statement on physical activity and exercise for cystic fibrosis: methodology and results of an international, multidisciplinary, evidence-driven expert consensus. Chron Respir Dis. 2022 Jan-Dec;19:14799731221121670. doi: 10.1177/14799731221121670. PMID 36068015
- [Background] Hebestreit H, Kieser S, Junge S, Ballmann M, Hebestreit A, Schindler C, Schenk T, Posselt HG, Kriemler S. Long-term effects of a partially supervised conditioning programme in cystic fibrosis. Eur Respir J. 2010 Mar;35(3):578-83. doi: 10.1183/09031936.00062409. Epub 2009 Jul 30. PMID 19643946
- [Background] Dwyer TJ, Alison JA, McKeough ZJ, Daviskas E, Bye PTP. Effects of exercise on respiratory flow and sputum properties in patients with cystic fibrosis. Chest. 2011 Apr;139(4):870-877. doi: 10.1378/chest.10-1158. Epub 2010 Sep 9. PMID 20829339
- [Background] Tejero Garcia S, Giraldez Sanchez MA, Cejudo P, Quintana Gallego E, Dapena J, Garcia Jimenez R, Cano Luis P, Gomez de Terreros I. Bone health, daily physical activity, and exercise tolerance in patients with cystic fibrosis. Chest. 2011 Aug;140(2):475-481. doi: 10.1378/chest.10-1508. Epub 2011 Feb 3. PMID 21292759
- [Background] Prevotat A, Godin J, Bernard H, Perez T, Le Rouzic O, Wallaert B. Improvement in body composition following a supervised exercise-training program of adult patients with cystic fibrosis. Respir Med Res. 2019 May;75:5-9. doi: 10.1016/j.resmer.2019.04.001. Epub 2019 Apr 13. PMID 31235455
- [Background] van de Weert-van Leeuwen PB, Hulzebos HJ, Werkman MS, Michel S, Vijftigschild LA, van Meegen MA, van der Ent CK, Beekman JM, Arets HG. Chronic inflammation and infection associate with a lower exercise training response in cystic fibrosis adolescents. Respir Med. 2014 Mar;108(3):445-52. doi: 10.1016/j.rmed.2013.08.012. Epub 2013 Aug 28. PMID 24480322
- [Background] Burtin C, Hebestreit H. Rehabilitation in patients with chronic respiratory disease other than chronic obstructive pulmonary disease: exercise and physical activity interventions in cystic fibrosis and non-cystic fibrosis bronchiectasis. Respiration. 2015;89(3):181-9. doi: 10.1159/000375170. Epub 2015 Feb 12. PMID 25676797
- [Background] Nixon PA, Orenstein DM, Kelsey SF, Doershuk CF. The prognostic value of exercise testing in patients with cystic fibrosis. N Engl J Med. 1992 Dec 17;327(25):1785-8. doi: 10.1056/NEJM199212173272504. PMID 1435933
- [Background] Saynor ZL, Gruet M, Rodriguez-Miguelez P, Harris RA. Oxygen transport and utilisation during exercise in cystic fibrosis: contributors to exercise intolerance. Exp Physiol. 2020 Dec;105(12):1979-1983. doi: 10.1113/EP088106. Epub 2020 Nov 11. PMID 33119143
- [Background] Cantin AM, Hartl D, Konstan MW, Chmiel JF. Inflammation in cystic fibrosis lung disease: Pathogenesis and therapy. J Cyst Fibros. 2015 Jul;14(4):419-30. doi: 10.1016/j.jcf.2015.03.003. Epub 2015 Mar 23. PMID 25814049
- [Background] Gruber W, Orenstein DM, Braumann KM, Beneke R. Interval exercise training in cystic fibrosis -- effects on exercise capacity in severely affected adults. J Cyst Fibros. 2014 Jan;13(1):86-91. doi: 10.1016/j.jcf.2013.06.005. Epub 2013 Jul 15. PMID 23863518
- [Background] Gao M, Huang Y, Wang Q, Liu K, Sun G. Effects of High-Intensity Interval Training on Pulmonary Function and Exercise Capacity in Individuals with Chronic Obstructive Pulmonary Disease: A Meta-Analysis and Systematic Review. Adv Ther. 2022 Jan;39(1):94-116. doi: 10.1007/s12325-021-01920-6. Epub 2021 Nov 18. PMID 34792785
- [Background] Jonas S, Izaurralde E. Towards a molecular understanding of microRNA-mediated gene silencing. Nat Rev Genet. 2015 Jul;16(7):421-33. doi: 10.1038/nrg3965. Epub 2015 Jun 16. PMID 26077373
- [Background] Ideozu JE, Zhang X, Rangaraj V, McColley S, Levy H. Microarray profiling identifies extracellular circulating miRNAs dysregulated in cystic fibrosis. Sci Rep. 2019 Oct 29;9(1):15483. doi: 10.1038/s41598-019-51890-7. PMID 31664087
- [Background] Catellani C, Cirillo F, Graziano S, Montanini L, Marmiroli N, Gulli M, Street ME. MicroRNA global profiling in cystic fibrosis cell lines reveals dysregulated pathways related with inflammation, cancer, growth, glucose and lipid metabolism, and fertility: an exploratory study. Acta Biomed. 2022 Jul 1;93(3):e2022133. doi: 10.23750/abm.v93i3.12842. PMID 35775757
- [Background] Dekkers JF, Wiegerinck CL, de Jonge HR, Bronsveld I, Janssens HM, de Winter-de Groot KM, Brandsma AM, de Jong NW, Bijvelds MJ, Scholte BJ, Nieuwenhuis EE, van den Brink S, Clevers H, van der Ent CK, Middendorp S, Beekman JM. A functional CFTR assay using primary cystic fibrosis intestinal organoids. Nat Med. 2013 Jul;19(7):939-45. doi: 10.1038/nm.3201. Epub 2013 Jun 2. PMID 23727931
- [Background] Bene Z, Fejes Z, Szanto TG, Fenyvesi F, Varadi J, Clarke LA, Panyi G, Macek M Jr, Amaral MD, Balogh I, Nagy B Jr. Enhanced Expression of Human Epididymis Protein 4 (HE4) Reflecting Pro-Inflammatory Status Is Regulated by CFTR in Cystic Fibrosis Bronchial Epithelial Cells. Front Pharmacol. 2021 May 14;12:592184. doi: 10.3389/fphar.2021.592184. eCollection 2021. PMID 34054511
- [Background] Fontes G, Ghislain J, Benterki I, Zarrouki B, Trudel D, Berthiaume Y, Poitout V. The DeltaF508 Mutation in the Cystic Fibrosis Transmembrane Conductance Regulator Is Associated With Progressive Insulin Resistance and Decreased Functional beta-Cell Mass in Mice. Diabetes. 2015 Dec;64(12):4112-22. doi: 10.2337/db14-0810. Epub 2015 Aug 17. PMID 26283735
- [Background] Plebani R, Potla R, Soong M, Bai H, Izadifar Z, Jiang A, Travis RN, Belgur C, Dinis A, Cartwright MJ, Prantil-Baun R, Jolly P, Gilpin SE, Romano M, Ingber DE. Modeling pulmonary cystic fibrosis in a human lung airway-on-a-chip. J Cyst Fibros. 2022 Jul;21(4):606-615. doi: 10.1016/j.jcf.2021.10.004. Epub 2021 Nov 17. PMID 34799298
- [Background] Fiz JA, Montserrat JM, Picado C, Plaza V, Agusti-Vidal A. How many manoeuvres should be done to measure maximal inspiratory mouth pressure in patients with chronic airflow obstruction? Thorax. 1989 May;44(5):419-21. doi: 10.1136/thx.44.5.419. PMID 2763242
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Murillo AMM, Tome-Amat J, Ramirez Y, Garrido-Arandia M, Valle LG, Hernandez-Ramirez G, Tramarin L, Herreros P, Santamaria B, Diaz-Perales A, Holgado M. Developing an Optical Interferometric Detection Method based biosensor for detecting specific SARS-CoV-2 immunoglobulins in Serum and Saliva, and their corresponding ELISA correlation. Sens Actuators B Chem. 2021 Oct 15;345:130394. doi: 10.1016/j.snb.2021.130394. Epub 2021 Jul 3. PMID 34248283
- [Background] Donadio MVF, Cobo-Vicente F, San Juan AF, Sanz-Santiago V, Fernandez-Luna A, Iturriaga T, Villa Asensi JR, Perez-Ruiz M. Is exercise and electrostimulation effective in improving muscle strength and cardiorespiratory fitness in children with cystic fibrosis and mild-to-moderate pulmonary impairment?: Randomized controlled trial. Respir Med. 2022 May;196:106798. doi: 10.1016/j.rmed.2022.106798. Epub 2022 Mar 1. PMID 35306386
- [Result] Divangahi M, Balghi H, Danialou G, Comtois AS, Demoule A, Ernest S, Haston C, Robert R, Hanrahan JW, Radzioch D, Petrof BJ. Lack of CFTR in skeletal muscle predisposes to muscle wasting and diaphragm muscle pump failure in cystic fibrosis mice. PLoS Genet. 2009 Jul;5(7):e1000586. doi: 10.1371/journal.pgen.1000586. Epub 2009 Jul 31. PMID 19649303
- [Result] King JA, Nichols AL, Bentley S, Carr SB, Davies JC. An Update on CFTR Modulators as New Therapies for Cystic Fibrosis. Paediatr Drugs. 2022 Jul;24(4):321-333. doi: 10.1007/s40272-022-00509-y. Epub 2022 May 16. PMID 35570261
- [Result] Rodriguez-Miguelez P, Seigler N, Ishii H, Crandall R, McKie KT, Forseen C, Harris RA. Exercise Intolerance in Cystic Fibrosis: Importance of Skeletal Muscle. Med Sci Sports Exerc. 2021 Apr 1;53(4):684-693. doi: 10.1249/MSS.0000000000002521. PMID 33105385
- [Result] Wells GD, Wilkes DL, Schneiderman JE, Rayner T, Elmi M, Selvadurai H, Dell SD, Noseworthy MD, Ratjen F, Tein I, Coates AL. Skeletal muscle metabolism in cystic fibrosis and primary ciliary dyskinesia. Pediatr Res. 2011 Jan;69(1):40-5. doi: 10.1203/PDR.0b013e3181fff35f. PMID 20938370
- [Result] Bene Z, Fejes Z, Macek M Jr, Amaral MD, Balogh I, Nagy B Jr. Laboratory biomarkers for lung disease severity and progression in cystic fibrosis. Clin Chim Acta. 2020 Sep;508:277-286. doi: 10.1016/j.cca.2020.05.015. Epub 2020 May 16. PMID 32428503
- [Result] Stachowiak Z, Wojsyk-Banaszak I, Jonczyk-Potoczna K, Narozna B, Langwinski W, Szczepankiewicz A. Extracellular vesicles-derived miRNAs as mediators of pulmonary exacerbation in pediatric cystic fibrosis. J Breath Res. 2023 Feb 10;17(2). doi: 10.1088/1752-7163/acb792. PMID 36720158
- [Derived] Pantoja-Arevalo L, Yvert T, Iturriaga T, Sanz-Santiago V, Barcelo O, Quesada-Gonzalez C, Morales-Tirado A, Santiago-Dorrego C, Lopez-Neyra A, Ruiz de Valbuena M, De Manuel Gomez C, Rubio Alonso M, De Vidania S, Ramirez-Castillejo C, Gonzalez-Gross M, Perez-Ruiz M. Strength-Oriented Virtual Exercise Training Intervention in Children and Adolescents with Cystic Fibrosis Under CFTR Modulators (the FIQMODE Study): Study Protocol for a Randomized Controlled Trial. Curr Protoc. 2025 Sep;5(9):e70202. doi: 10.1002/cpz1.70202. PMID 40966068